CLINICAL TRIAL: NCT03902119
Title: Effectiveness of a New Tool (INYBI) in Individuals With Chronic Non-specific Neck Pain.
Brief Title: INYBI Tool in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, Assistant Proffesor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INYBI tool
Record Dates: First submitted 2019-03-27; First posted 2019-04-03 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Neck Pain
Keywords: neck pain; randomized control trial; manual therapy; physical therapy; suboccipital inhibition
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INIBY tool (Experimental): Patients will undergo a single treatment session consisting of applying a suboccipital muscle inhibition technique using the so-called INYBI tool. The treatment session will last approximately 5 minutes
  Interventions: Device: INYBI tool
- Manual suboccipital inhibition (Active Comparator): Patients will receive a single treatment session consisting of the use of the manual suboccipital muscles inhibition technique.The treatment session will last approximately 5 minutes
  Interventions: Other: Manual suboccipital inhibition

INTERVENTIONS:
Device: INYBI tool — Patients will lie down in supine position so that the INYBI tool will contact the suboccipital muscles at the posterior arch of the atlas. The therapist will adapt the height of the tool for each individual. All patients will use the softest head of the device. A 50Hz vibration speed will be set sup during 5 minutes.
  Arms: INIBY tool
Other: Manual suboccipital inhibition — Patients will lie down in supine position.The therapist will be seated at the head of the treatment table. The therapist will keep the metacarpophalangeal joints in a flexed position, while therapists fingertips of both hands will contact with the suboccipital muscles at the posterior arch of the atlas.
  Arms: Manual suboccipital inhibition

SUMMARY:
Objectives: To evaluate the clinical efficacy of using a manual inhibition technique for the suboccipital muscles compared with the use of the so-called INYBI tool in individuals with chronic non-specific neck pain, and the compare the results of using both approaches on pain relief, cervical range of motion neck and vertical maximum mouth opening.

Design: Quantitative, experimental, longitudinal, prospective, and double blinded study.

Subjects: Patients between 18 and 40 years, with chronic non-specific neck pain of at least 3 months of evolution.

Methods: The experimental group will undergo a 5 minutes intervention for the suboccipital muscles using the INYBI tool. The control group will receive a 5 minutes of treatment involving the suboccipital muscles manual inhibition technique.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-specific mechanical neck pain.
* Pain of more than 3 months of duration.
* Pain between the occiput and the third dorsal vertebra.
* Willingness to participate in the treatment and in the follow-up measurements
* Neck pain reproduced by neck movements or palpation

Exclusion Criteria:

* Cognitive impairment or inability to communicate.
* Having received manual therapy in the last two months before recruitment.
* Having received anti-inflammatory treatment, antidepressants or muscle relaxants in the last 72 hours.
* Any contraindication to treatment or evaluation procedures.
* Diagnosis of systemic diseases
* Diagnosis of fibromyalgia
* Pregnancy
* Signs of spinal nerve root compression
* Previous whiplash
* Any diagnosed possible cause for their neck pain (infection, cancer, spinal stenosis)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) in the evaluated muscles. The PPT levels will be evaluated in Kilograms / cm2 | From baseline to immediately after treatment.
  PPT levels, defined as the minimum necessary pressure to evoke pain will be evaluated using a handheld electronic pressure algometer.
Active cervical range of movement (ROM). The range of movement will be assessed in degrees | From baseline to immediately after treatment.
  Flexion, extension, left and right side flexion, and left and right rotation will be assessed using a digital inclinometer.
Pain free vertical mouth opening. This outcome will be evaluated in centimeters. | From baseline to immediately after treatment.
  Maximum pain free vertical mouth opening will be assessed using a digital caliper that will place between the incisors 11, 21, 31 y 41.
Atlas rotation ROM, assessed in degrees | From baseline to immediately after treatment.
  The atlas bone left and right rotation ROM will be assessed using the flexion-rotation test. For this test, with the participant in supine position, the maximum mobility in head rotation while keeping maximum passive neck flexion will be assessed
Self-reported pain intensity | From baseline to immediately after treatment.
  Self-perceived pain intensity will be evaluated during all active cervical movements by a 0 to 10 Visual Analogue Scale (VAS), where 0 denotes no pain at all, and 10 denotes the maximum possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Heredia-Rizo, PhD, Study Director — Physiotherapy Department, University of Sevilla, Spain
Locations (1):
- University of Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No